CLINICAL TRIAL: NCT02259855
Title: Open Label, Study to Determine the Pharmacokinetic Interactions of Steady State Tipranavir/Ritonavir (500/200 mg) and Steady State Ribavirin and Pegylated Interferon Alfa 2a in HIV Negative, HCV Infected Subjects With Mild Hepatic Impairment and the Pharmacokinetic Properties of Tipranavir/Ritonavir in HIV Negative, HCV, HBV, Hepatitis Delta Infected Subjects or Alcoholic Cirrhosis Subjects With Moderate Hepatic Impairment
Brief Title: Pharmacokinetics (PK) of Tipranavir/Ritonavir, Ribavirin, Pegylated Interferon (Peg INF) in Hepatitis C (HCV) Subjects With Mild Hepatic Impairment and in HCV, Hepatitis B (HBV), Hepatitis D Infected Subjects or Alcoholic Cirrhosis With Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1182.59
Record Dates: First submitted 2014-09-24; First posted 2014-10-09 (Estimated); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — tipranavir; Ritonavir; Ribavirin

STUDY DESIGN:
Oversight: FDA-regulated Device: No

ARMS (3):
- Mild hepatic insufficiency (Experimental)
  Interventions: Drug: Tipranavir; Drug: Ritonavir; Drug: Pegylated interferon; Drug: Ribavirin
- Moderate hepatic insufficiency (Experimental)
  Interventions: Drug: Tipranavir; Drug: Ritonavir
- Healthy subjects (Experimental)
  Interventions: Drug: Tipranavir; Drug: Ritonavir

INTERVENTIONS:
Drug: Tipranavir
Drug: Ritonavir
Drug: Pegylated interferon
  Arms: Mild hepatic insufficiency
Drug: Ribavirin
  Arms: Mild hepatic insufficiency

SUMMARY:
The primary objectives were:

* To determine the effects of steady state TPV co-administered with low dose RTV on steady state PegIFN and RBV in HIV negative subjects with mild hepatic impairment (scheme A)
* To determine the effects of steady state of pegylated interferon (PegIFN) and RBV on steady state pharmacokinetics of TPV co-administered with low dose RTV in HIV negative subjects with mild hepatic impairment (scheme A)
* To determine the pharmacokinetics of single dose and steady state TPV/r 500/200 mg in subjects with moderate hepatic insufficiency (scheme B)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and Age ≤ 75 years
* BMI ≥18 and BMI ≤ 29 kg/m2 (Body Mass Index) at screening visit
* Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and the local legislation
* Ability to swallow multiple large capsules without difficulty
* Serologic evidence of chronic hepatitis C infection by an antibody test and HCV branched DNA (bDNA) for subjects with mild hepatic impairment (Scheme A)
* Serologic evidence of chronic hepatitis C, B and/or delta infection by an antibody test and HCV bDNA, HBV RNA polymerase chain reaction (PCR) for subjects with moderate hepatic impairment (Child Pugh B)
* Alcoholic cirrhosis, for subjects with moderate hepatic impairment (Child Pugh B). Patients had to stop the alcohol consumption at least 1 month before the screening without any evidence of acute alcoholic hepatitis
* Subjects HCV positive with mild hepatic insufficiency were to be on stable treatment with PegIFN and ribavirin since at least 12 weeks prior to study entry
* Subjects with mild hepatic insufficiency were to be viral non-responders with less than a 2 log reduction in HCV RNA, compared to baseline (HCV treatment initiation) and have positive HCV RNA after 12 weeks therapy with PegIFN/RBV
* Subjects with:

  * stable mild hepatic insufficiency treated by PegIFN and RBV
  * moderate hepatic insufficiency [Child-Pugh Class B (score 7-9)]
* All fertile males or females, and their respective partner(s) were to be using two forms of effective contraception during ribavirin treatment and during the 6 months after its end. All other women must agree to use an effective form of contraception during the entire duration of the study. This may include condoms, diaphragms or implants. This did not apply to those surgically sterilized or in a post menopausal state
* Laboratory values that indicated adequate baseline organ function were required at the time of screening. All subjects with mild and moderate hepatic insufficiency should have all laboratory values less than or equal to grade 2, based on division of aids (DAIDS) Grading Scale. The following exceptions were made:

  * Alanine transaminase (ALT) and/or aspartate aminotransferase (AST) < 3 x upper limit of normal (ULN)
  * Alkaline Phosphatase < 2 x ULN
  * Haemoglobin > 10.0 g/dL
  * Platelets > 50.000 / μl And all healthy control subjects should have all laboratory values < grade 1
* Willingness to abstain from alcohol starting 2 days prior to administration of study drug up to the end of the study, to abstain from over counter herbal medications for the duration of the trial
* Willingness to abstain from the following starting 14 days prior to administration of study medication up until the end of the study: Grapefruit or grapefruit juice, red wine, seville oranges (marmalade), St John's Wort or Milk Thistle
* Willingness to abstain from the following 72 h prior to PK sampling: Garlic supplements, Methylxanthine containing drinks (coffee, tea, cola, energy drinks, chocolate, etc.)
* Acceptable medical history, physical examination were required prior to entering the treatment phase of the trial
* Reasonable probability for completion of the study, including dosing requirements of TPV/r and acceptance of the risk for hepatic decompensation

Exclusion Criteria:

* Use of any medication listed in the protocol within 30 days prior to Day 1
* Participation in another trial with an investigational medicine within 2 months prior to Day 1
* Absolute neutrophil count (ANC) < 750 cells/mm³ at screening
* Serum creatine level > 1.5 times upper the limit of normal at screening
* History of acute illness within 60 days prior to Day 1
* Subject with mild hepatic impairment (scheme A), HIV, HBV, hepatitis Delta positive and/or alcoholic cirrhosis
* Subject with moderate hepatic impairment (CPB), HIV positive
* Subject control, HIV hepatitis positive and alcoholic cirrhosis
* Subjects HIV positive, HBV positive and, for subjects controls HCV positive
* Active bleeding from oesophageal varices or other conditions consistent with active decompensated liver disease, active spontaneous bacterial peritonitis, active oesophageal variceal disease or active liver encephalopathy
* Subjects with Child-Pugh Class C (score > 9)
* Alcohol abuse within 1 month prior to screening or during the study
* Other substance abuse within 6 months prior to screening or during the study
* Subjects with a history of any illness or allergy (including drug allergy) that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering TPV and RTV
* Subjects who have taken (within 7 days prior to Day 1) any over-the-counter or prescription medication that, in the opinion of the investigator in consultation with the Boehringer Ingelheim France (BIF) clinical monitor, might interfere with absorption, distribution, or metabolism of the study medications
* Known hypersensitivity to sulphonamide class of drugs
* Known hypersensitivity to TPV, RTV or antiretroviral drugs (marketed or experimental use as part of clinical research studies)
* Known elevated liver enzymes in past clinical trials with any compounds
* Inability to adhere to the protocol
* Cautions or warnings in the RTV, PegIFN and RBV package insert which, in the opinion of the investigator, constituted grounds for subject exclusion
* History or other evidence of severe illness, malignancy or any other conditions which would have made the patients, in the opinion of the investigator, unsuitable for the trial
* History of any systemic antineoplasic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) ≤ 6 months prior to study entry or expectation that such treatment would be needed at any time during the study
* Use of hormone replacement therapy with oestrogen-based preparations for at least 1 month prior to screening and for the duration of the study
* Administration of antimicrobial agents within 10 days prior to Day 1 (Visit 2)
* Subjects with evidence of hepatocellular carcinoma, or who tested positive for serum alpha foeto protein > 5μg/l or suspected tumour based on ultrasonography examination, - Patients with history of stroke, intracranial aneurysm, neurosurgery and skull traumatism within 4 weeks prior to screening
* History of intracranial, intraocular, spinal, retroperitoneal or atraumatic intraarticular bleeding
* Gastrointestinal hemorrhage within the past year
* Endoscopically documented gastro-duodenal ulcer disease in the previous 30 days
* Hemorrhagic disorder or bleeding diathesis
* Need for anticoagulant treatment for disorders
* Uncontrolled hypertension (systolic blood pressure (SBP) >180 mmHg and/or diastolic blood pressure (DBP) >100 mmHg)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2008-10-01 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from 0 to 12 hours of ribavirin (RBV), tipranavir (TPV) and ritonavir (RTV) in the plasma (AUC0-12h) | Pre-dose, up to 120 hours after start of treatment
Area under the concentration-time curve from 0 to 24 hours of pegylated interferon (Peg IFN) in the plasma (AUC0-24h) | Pre-dose, up to 120 hours after start of treatment
Maximum measured concentration of RBV, Peg INF, TPV and RTV in the plasma (Cmax) | Pre-dose, up to 120 hours after start of treatment
Measured concentration of RBV, TPV and RTV in the plasma at 12 hours (Cp12h) | Pre-dose, up to 120 hours after start of treatment
Measured concentration of Peg INF in the plasma at 24 hours (Cp24h) | Pre-dose, up to 120 hours after start of treatment
Area under the concentration-time curve from 0 extrapolated to infinity of TPV and RTV in the plasma (AUC0-∞) | Pre-dose, up to 120 hours after start of treatment

SECONDARY OUTCOMES:
Time from dosing to the maximum concentration of the analytes in the plasma (tmax) | Pre-dose, up to 120 hours after start of treatment
Terminal half-life of the analytes in the plasma (t1/2) | Pre-dose, up to 120 hours after start of treatment
Apparent clearance of the analytes in the plasma after extra vascular administration (CL/F) | Pre-dose, up to 120 hours after start of treatment
Apparent volume of distribution of the analytes in the plasma (Vz/F) | Pre-dose, up to 120 hours after start of treatment
Number of patients with clinically significant changes in laboratory values | up to 3 weeks after start of treatment
Number of patients with adverse events | Up to 7 weeks
Number of patients with clinically significant changes in vital signs (seated blood pressure, pulse rate) | up to 3 weeks after start of treatment
Number of patients with clinically significant changes from baseline in 12-lead ECG | 3 weeks after start of treatment
Assessment of tolerability by the investigator | Up to 3 weeks after start of treatment
  verbal rating scale

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com